CLINICAL TRIAL: NCT02056665
Title: Randomized Clinical Trial, Placebo Compared to Evaluate the Efficacy and Safety of Minocycline in Angelman Syndrome
Brief Title: Study to Evaluate the Efficacy and Safety of Minocycline in Angelman Syndrome
Acronym: A-MANECE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Puerta de Hierro University Hospital (Other)
Responsible Party: Principal Investigator, BELEN RUIZ-ANTORAN, DR, Puerta de Hierro University Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A-MANECE
Record Dates: First submitted 2014-02-05; First posted 2014-02-06 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Angelman Syndrome
Keywords: Angelman Syndrome; EFFICACY; SAFETY; MINOCYCLINE; Pediatrics population; Rare diseases
MeSH Terms: conditions — Angelman Syndrome; cyclopia sequence; Rare Diseases | interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- MINOCYCLINE 8 weeks (Experimental): Duration of treatment: 8 weeks
  * Patients <35 kg. 100 mg / day. Administered at a dose of one capsule of 50 mg breakfast and dinner.
  * Patients 35 - 50 kg. 150 mg / day. Administered at a dose of 2 capsules of 50 mg breakfast and 1 capsule of 50mg dinner.
  * Patients > 50 kg. 200 mg / day. Administered at a dose of two capsules of 50 mg of breakfast and dinner.
  Interventions: Drug: MINOCYCLINE; Drug: PLACEBO (for Minocycline)
- PLACEBO 8 weeks (Placebo Comparator): Pill manufactured to mimic Minocycline 50 mg capsule
  Interventions: Drug: MINOCYCLINE; Drug: PLACEBO (for Minocycline)
- MINOCYCLINE 16 weeks (Experimental): Duration of treatment: 16 weeks
  Patients <35 kg. 100 mg / day. Administered at a dose of one capsule of 50 mg breakfast and dinner.
  Patients 35 - 50 kg. 150 mg / day. Administered at a dose of 2 capsules of 50 mg breakfast and 1 capsule of 50mg dinner.
  Patients > 50 kg. 200 mg / day. Administered at a dose of two capsules of 50 mg of breakfast and dinner.
  Interventions: Drug: MINOCYCLINE

INTERVENTIONS:
Drug: MINOCYCLINE — Pill Minocycline 50 mg capsule
  Other Names: Commercial name: Aknemin 50; Active substance: MINOCYCLINE; Administration routes: Oral use
Drug: PLACEBO (for Minocycline) — Pill manufactured to mimic Minocycline 50 mg capsule
  Other Names: Commercial name: NA; Non Active substance:; Administration routes: Oral use
  Arms: MINOCYCLINE 8 weeks; PLACEBO 8 weeks

SUMMARY:
RANDOMIZED CLINICAL TRIAL, PLACEBO COMPARED TO EVALUATE THE EFFICACY AND SAFETY OF MINOCYCLINE IN ANGELMAN SYNDROME (A-MANECE STUDY)

DETAILED DESCRIPTION:
STUDY TO EVALUATE THE EFFICACY AND SAFETY OF MINOCYCLINE IN ANGELMAN SYNDROME

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 6 and 30 years old.
* Clinical diagnosis of Angelman Syndrome and molecular confirmation of diagnosis.
* The participant has an acceptable guardian can give consent on behalf of the participant.

Exclusion Criteria:

* Patients with hypersensitivity to tetracyclines.
* Patients with impaired hepatic or renal function and in those with mainly drug allergy history.
* Any other condition that in the opinion of the investigator is considered clinically relevant and that administration of minocycline contraindicated

Ages: 6 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2014-01; Primary Completion 2014-09 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Increased on the equivalent age of development | 8, 16 and 24 weeks
  Increased on the equivalent age of development, obtained through Development Scale R Merrill-Palmer (MP-R)

SECONDARY OUTCOMES:
Improved specific cognitive, language and communication, motor development, social-emotional and adaptive behavior | 8, 16 and 24 weeks
  Improved specific cognitive, language and communication, motor development, social-emotional and adaptive behavior obtained through Development Scale R Merrill-Palmer (MP-R)
Improvement of EEG. | 8, 16 and 24 weeks
  Improvement of EEG. Measure based on changes in the background activity, type, number and duration of crises, widespread tendency to crises, paroxysmal abnormalities recorded types and the overall evaluation of clinical neurophysiologist
Safety and tolerability | 8, 16 and 24 weeks
  a) Physical Examination b) Vital signs c) Laboratory Tests d) Adverse effects (AEs) list for treatment, laboratory values, values outside the reference range and descriptive statistics.
Clinical Global impression (CGI) | 8, 16 and 24 weeks
  Improvement of CGI. . Measure based on changes in the Clinical Global Impression through the perception of parents or guardians, you neurologists and therapist

CONTACTS AND LOCATIONS:
Overall Officials: Belen Ruiz-Antorán, Principal Investigator — Clinical Pharmacology. Puerta de Hierro University Hospital
Locations (1):
- Puerta de Hierro University Hospital, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Ruiz-Antoran B, Sancho-Lopez A, Cazorla-Calleja R, Lopez-Pajaro LF, Leiva A, Iglesias-Escalera G, Marin-Serrano ME, Rincon-Ortega M, Lara-Herguedas J, Rossignoli-Palomeque T, Valiente-Rodriguez S, Gonzalez-Marques J, Roman-Riechmann E, Avendano-Sola C. A randomized placebo controlled clinical trial to evaluate the efficacy and safety of minocycline in patients with Angelman syndrome (A-MANECE study). Orphanet J Rare Dis. 2018 Aug 20;13(1):144. doi: 10.1186/s13023-018-0891-6. PMID 30126448